CLINICAL TRIAL: NCT02222597
Title: An Evaluation of Near-Infrared Spectroscopy for Intracranial Hematoma Detection of Head Trauma Patients in the Emergency Department.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201209046DPB
Record Dates: First submitted 2014-08-20; First posted 2014-08-21 (Estimated); Last update posted 2014-08-26 (Estimated); Status verified 2014-08

CONDITIONS: Within 12 Hrs of Head Injury
Keywords: head injury; infrascanner; intracranial hemorrhage
MeSH Terms: conditions — Craniocerebral Trauma; Intracranial Hemorrhages

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- positive infrascanner finding
  Interventions: Device: infrascanner

INTERVENTIONS:
Device: infrascanner

SUMMARY:
The purpose of this study is to evaluate Near-Infrared Spectroscopy for intracranial hematoma detection of head trauma patients

ELIGIBILITY:
Inclusion Criteria:

The patients within 12 hours after head injury, visiting the Emergency Department of the National Taiwan University Hospital, and receiving computed tomography of head were enrolled.

Exclusion Criteria:

1. The patients over 12 hours after head injury, visiting the Emergency Department of the NTUH, and receiving computed tomography of head were excluded.
2. Patients with massive scalp laceration or hematoma were excluded. -

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The patients within 12 hours after head injury visit the Emergency Department of the NTUH.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2014-04; Primary Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
detect the predictive value of the infrascanner for intracranial hemorrhage | within 12 hours after head injury

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital Emergency Department, Taipei, Taiwan, Taiwan